CLINICAL TRIAL: NCT04900311
Title: Pyrotinib Versus Pertuzumab in Combination With Neoadjuvant Trastuzumab and Nab-Paclitaxel in HER2+ Early or Locally Advanced Breast Cancer
Acronym: Pyramid
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-020
Record Dates: First submitted 2021-04-28; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-04

CONDITIONS: HER2+ Early or Locally Advanced Breast Cancer
Keywords: HER2+ breast cancer; neoadjuvant; pyrotinib
MeSH Terms: interventions — pyrotinib; Trastuzumab; 130-nm albumin-bound paclitaxel; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- pyrotinib + trastuzumab + nab-paclitaxel (Experimental)
  Interventions: Drug: pyrotinib + trastuzumab + nab-paclitaxel
- pertuzumab + trastuzumab + nab-paclitaxel (Active Comparator)
  Interventions: Drug: pertuzumab + trastuzumab + nab-paclitaxel

INTERVENTIONS:
Drug: pyrotinib + trastuzumab + nab-paclitaxel — patients will be treated every 3 weeks for four cycles prior to surgery at following doses: pyrotinib: 400 mg/day, orally, qd trastuzumab: IV infusion on Day 1 every 3 weeks with loading dose of 8 mg/kg in Cycle 1, and 6 mg/kg in Cycles 2-4 nab-paclitaxel: 260 mg/m2 IV infusion on Day 1 every 3 weeks, or 125 mg/m2 IV infusion on Days 1, 8 and 15 every 3 weeks (the nab-paclitaxel administration cycle was determined by investigator at each site)
  Arms: pyrotinib + trastuzumab + nab-paclitaxel
Drug: pertuzumab + trastuzumab + nab-paclitaxel — patients will be treated every 3 weeks for four cycles prior to surgery at following doses: pertuzumab: IV infusion on Day 1 every 3 weeks with loading dose of 840 mg for Cycle 1, followed by 420 mg for Cycles 2-4 trastuzumab: IV infusion on Day 1 every 3 weeks with loading dose of 8 mg/kg in Cycle 1, and 6 mg/kg in Cycles 2-4 nab-paclitaxel: 260 mg/m2 IV infusion on Day 1 every 3 weeks, or 125 mg/m2 IV infusion on Days 1, 8 and 15 every 3 weeks (the nab-paclitaxel administration cycle was determined by investigator at each site)
  Arms: pertuzumab + trastuzumab + nab-paclitaxel

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of pyrotinib versus pertuzumab in combination with trastuzumab and nab-paclitaxel for neoadjuvant treatment in HER2+ early or locally advanced breast cancer patients. To explore whether pyrotinib regimen could provide better clinical results compared with pertuzumab in the study population.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, open-label, controlled trial. Eligible patients will be randomized to neoadjuvant pyrotinib or pertuzumab containing regimen every 3 weeks for four cycles before surgery. Randomization was stratified by the following factors: hormone receptor status and primary tumor size. After completing four cycles of neoadjuvant treatment, all patients who are eligible for surgery will undergo surgery and have their pathologic response evaluated. Following surgery, patients will receive 90-100 mg/m2 epirubicin and 600 mg/m2 cyclophosphamide every 3 weeks for 4 cycles. Clinicians will select subsequent treatments for patients based on guidelines as well as clinical practice at each site.

ELIGIBILITY:
Inclusion Criteria:

* female patients, treatment-naïve, aged ≥ 18 years and ≤ 75 years;
* ECOG score 0-1 (ECOG, Eastern Cooperative Oncology Group);
* Histologically confirmed invasive breast cancer (early stage or locally advanced) :Primary tumor greater than 2 cm diameter and cT2-cT4/cN0-cN3/cM0 (clinical stage II and III);
* HER2 expression positive breast cancer confirmed by pathological examination,
* known hormone receptor status (ER and PR);
* the level of major organ function must meet the following requirements: blood routine test: neutrophil (ANC) ≥ 1.5 × 109/L; platelet count (PLT) ≥ 90 × 109/L; hemoglobin (Hb) ≥ 90g/L; blood biochemistry test: total bilirubin (TBIL) ≤ 2.5 × ULN (upper normal limit); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 × ULN; alkaline phosphatase ≤ 2.5 × ULN; blood urea nitrogen (BUN) and creatinine (Cr) ≤ 1.5 × ULN; echocardiography: LVEF ((Left Ventricular Ejection Fraction) ≥ 55%; 12 ECG: QT interval corrected by Fridericia method (QTcF) < 470 ms in women
* Female subjects who have not yet experienced menopausal or not surgically sterile agree to practice abstinence or use effective methods of contraception for at least 7 months during and after the last dose of study drug;
* Sign the informed consent form and are willing to cooperate in the follow-up.

Exclusion Criteria:

* breast cancer of both sides, stage IV breast cancer or metastatic breast cancer;
* inflammatory breast cancer;
* History of other malignancy, or previous anti-cancer therapy or radiotherapy for any malignancy, excluding cured carcinoma in situ of the cervix or squamous or basal cell carcinoma.
* simultaneously participated in other clinical trials;
* Major surgical procedure unrelated to breast cancer within 4 weeks prior to randomization or from which the patient has not fully recovered
* blood transfusion, or received colony-stimulating factor treatments before randomization;
* known history of allergy to any of the study medications and any of the ingredients or excipients of these medications;
* history of immunodeficiency, including positive HIV test, or suffering from other acquired, congenital immunodeficiency diseases, or history of organ transplantation.
* had any heart disease, including: (1) angina pectoris; (2) arrhythmia that is clinically significant or required medication; (3) myocardial infarction; (4) heart failure; (5) any other heart disease judged by the investigator as not suitable for this trial.
* pregnant or lactating
* Other concurrent serious diseases that are serious hazards to the patient's safety or may interfere with planned treatment (including but not limited to hypertension, severe diabetes, active infection, thyroid disease, etc.) ;
* Inability to swallow, chronic diarrhea, bowel obstruction, and other factors affecting medication intake and absorption.
* Any other condition that, in the opinion of the investigator, makes the subject unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
tpCR (totally pathological Complete Response) assessed by the IRC(Independent Review Committee) | Pathologic response will be evaluated right after surgery, which will be performed within 14 days after the completion neoadjuvant therapy (four cycles, 21 days per cycle).
  defined as the absence of any residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes following completion of neoadjuvant therapy and surgery.

SECONDARY OUTCOMES:
iDFS (Invasive disease-free survival) | from the date of surgery till two years after study-defined treatment.
  iDFS, defined as the time from the first date of no disease (i.e., date of surgery) to the first documentation of one of the following events:
  1. Disease recurrence (local, regional, distant, or contralateral) after surgery
  2. Death from any cause
EFS (event free survival) | from the date of surgery till two years after study-defined treatment.
  EFS, defined as time from randomization to the first documentation of one of the following events:
  1. Disease progression (before surgery), as determined by the investigator using RECIST v1.1 Any evidence of in situ contralateral disease will not be identified as progressive disease (PD). Any evidence of invasive contralateral disease will be considered disease progression
  2. Disease recurrence (local, regional, distant, or contralateral) after surgery
  3. Death from any cause
ORR (Objective Response Rate) | At the end of neoadjuvant therapy (four cycles, 21 days per cycle).
  the proportion of patients who achieved Complete Response (CR) or Partial Response (PR) during Cycles 1-4, according to RECIST v1.1
the rate of adopting breast-conserving surgery | evaluated right after surgery, which will be performed within 14 days after the completion neoadjuvant therapy (four cycles, 21 days per cycle).
  the proportion of patients who have undergone breast-conserving surgery

OTHER OUTCOMES:
Incidence of serious adverse events and other adverse events of special interest | through study completion, an average of 2.5 years.
  Assess the incidence of serious adverse events (SAEs) and other adverse events.
Exploratory biomarker analyses | through study completion, an average of 2.5 years.
  The correlation between baseline molecular biomarkers and efficacy outcomes will be evaluated. Biomarkers may include blood lipids and metabolomics profiles based on Nuclear Magnetic Resonance techniques.